CLINICAL TRIAL: NCT03649477
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled, 8-week Clinical Study to Assess the Efficacy, Safety, and Tolerability, of Intranasal Carbetocin (LV-101) in Prader-Willi Syndrome (PWS) With Long Term Follow-Up (CARE-PWS)
Brief Title: Phase 3 Study of Intranasal Carbetocin (LV-101) in Patients With Prader-Willi Syndrome
Acronym: CARE-PWS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Levo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LV-101-3-01
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-08

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader-Willi syndrome; carbetocin
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Intervention Model Description: Three parallel groups (two different doses of carbetocin and placebo) for the first 8 weeks; two parallel groups (two different doses of carbetocin) during 56 weeks of follow-up and the optional extension period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): matched placebo during first 8-weeks; prospectively randomized 1:1 to either one of the two doses of carbetocin during 56-week follow-up and optional extension periods
  Interventions: Drug: placebo
- 3.2 mg of LV-101 (Experimental): 3.2 mg of LV-101 during first 8-weeks; remain on same dose during 56-week follow-up and optional extension periods
  Interventions: Drug: 3.2 mg intranasal carbetocin
- 9.6 mg of LV-101 (Experimental): 9.6 mg of LV-101 during first 8-weeks; remain on same dose during 56-week follow-up and optional extension periods
  Interventions: Drug: 9.6 mg intranasal carbetocin

INTERVENTIONS:
Drug: 3.2 mg intranasal carbetocin — three times per day with meals
  Other Names: LV-101
  Arms: 3.2 mg of LV-101
Drug: 9.6 mg intranasal carbetocin — three times per day with meals
  Other Names: LV-101
  Arms: 9.6 mg of LV-101
Drug: placebo — three times per day with meals
  Arms: Placebo

SUMMARY:
This Phase 3 study is designed to test the effectiveness of intranasal carbetocin (LV-101) in participants with Prader-Willi syndrome (PWS). Carbetocin is an oxytocin analog (a man-made chemical that is like oxytocin). This study will also evaluate the safety and tolerability of LV-101.

DETAILED DESCRIPTION:
This is a Phase 3 randomized, double-blind study with an 8-week, placebo-controlled period designed to test the effectiveness, safety, and tolerability of LV-101 in participants with PWS.

Effectiveness will be measured using both caregiver-reported and clinician-reported measures of hyperphagia (extreme hunger), obsessive and compulsive behaviors, and anxiety. Safety and tolerability will be measured by adverse events, laboratory tests, and physical exams.

After the 8-week placebo-controlled period, there will be a long-term follow-up period of 56 weeks and an optional extension period after study week 64 during which all participants will receive active treatment with LV-101. At Week 8, participants who were randomized to placebo in the placebo-controlled period will be randomized to one of the two LV-101 doses, administered three times per day before meals.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-confirmed Prader-Willi syndrome
* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of participant); provide voluntary, written assent (participants, as appropriate)
* PWS Nutritional Phase 3 (hyperphagic, rarely feels full)

Exclusion Criteria:

* Living in a group home
* Genetically diagnosed Schaaf-Yang syndrome or other genetic, hormonal, or chromosomal cognitive impairment
* New food-related interventions, including environment or dietary restrictions, within 1 month of screening
* Dose of any allowed chronic concomitant medications or supplements that have not been stable for ≥3 months prior to the study or is not expected to remain stable while participating in the study; adjustments in growth hormone dose ≤10% are not exclusionary
* Presence of cardiovascular disorders, epilepsy, frequent migraines, or severe asthma
* More than 3 episodes of sinusitis in the 12 months prior to Screening Visit or presence of nasal diseases that may affect deposition of intranasal medication
* Unwilling to abstain from nasal saline, other nasal irrigation, or other intranasal medications for 2 weeks prior to the Baseline visit and during the 8-week, placebo-controlled period of the study
* Use of weight loss medication, oxytocin, carbetocin, or vasopressin in the 6 months prior to screening
* Participation in an interventional research study involving another investigational medication or device in the 6 months prior to screening or during the study
* Based on the judgment of the Investigator, is unsuitable for the study for any reason, including but not limited to unstable medical condition, inability to comply with the protocol, or other risk to subject or to the integrity of the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2022-07-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles (USC), Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Harvard Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Tulsa, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Queensland Children's Hospital, South Brisbane, Queensland, Australia
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Toronto Hospital for Sick Kids, Toronto, Ontario
  - CHU Ste Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roof E, Deal CL, McCandless SE, Cowan RL, Miller JL, Hamilton JK, Roeder ER, McCormack SE, Roshan Lal TR, Abdul-Latif HD, Haqq AM, Obrynba KS, Torchen LC, Vidmar AP, Viskochil DH, Chanoine JP, Lam CKL, Pierce MJ, Williams LL, Bird LM, Butler MG, Jensen DE, Myers SE, Oatman OJ, Baskaran C, Chalmers LJ, Fu C, Alos N, McLean SD, Shah A, Whitman BY, Blumenstein BA, Leonard SF, Ernest JP, Cormier JW, Cotter SP, Ryman DC. Intranasal Carbetocin Reduces Hyperphagia, Anxiousness, and Distress in Prader-Willi Syndrome: CARE-PWS Phase 3 Trial. J Clin Endocrinol Metab. 2023 Jun 16;108(7):1696-1708. doi: 10.1210/clinem/dgad015. PMID 36633570

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in three countries, the United States, Canada and Australia. The first participant was screened in November 2018, the first participant was enrolled in December 2018, and the last participant was enrolled in March 2020.
Pre-assignment Details: Subjects were randomized 1:1:1 at Baseline to receive the 9.6 mg/dose, 3.2 mg/dose, or placebo during the 8-week placebo-controlled period. A total of 130 subjects were evaluated (44 subjects in the 9.6 mg/dose arm, and 43 subjects each in the 3.2 mg/dose and placebo arms). Of these 130 subjects, 128 subjects (98.5%) completed the Week 8 visit and entered into the long-term follow-up period.
Groups:
- 9.6 mg of LV-101: 9.6 mg of LV-101 during the 8-week placebo-controlled period
  9.6 mg intranasal carbetocin: three times per day with meals
- 3.2 mg of LV-101: 3.2 mg of LV-101 during the 8-week placebo controlled period
  3.2 mg intranasal carbetocin: three times per day with meals
- Placebo: Matched intranasal placebo during the 8-week placebo controlled period
  placebo: three times per day with meals
Period: Overall Study
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Started | 44 | 43 | 43
Completed | 42 | 43 | 43
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 43 | 130
Age, Categorical [Count of Participants; unit: Participants] — Inclusion criteria was 7 to 18 years of age at Screening. Subjects who were 19 years of age at Baseline were still eligible to participate if all other eligibility criteria were met.
  Participants
    <=18 years | 42 | 43 | 43 | 128
    Between 18 and 65 years | 2 | 0 | 0 | 2
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 27 | 24 | 72
  Male | 23 | 16 | 19 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 13
  Not Hispanic or Latino | 40 | 38 | 39 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 37 | 37 | 37 | 111
  More than one race | 3 | 2 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hyperphagia Behavior
Description: Change in hyperphagia (extreme hunger) as measured by the Hyperphagia Questionnaire for Clinical Trials (HQ-CT) Total Score versus placebo.
  Score range: 0-36; higher scores mean a worse outcome. Reduction in score indicates improvement.
Time Frame: Baseline to Week 8
Population: Primary Analysis Set: A subset of the Full Analysis Set that included all subjects with at least one post-Baseline visit (i.e., Week 2 or Week 8) completed prior to March 01, 2020 and excluded all efficacy data collected on or after March 01, 2020.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Number analyzed (Participants) | 40 | 39 | 40
score on a scale | -3.439 [-5.304 to -1.575] | -5.372 [-7.259 to -3.486] | -2.237 [-4.095 to -0.378]
Statistical Analysis 1: Comparison: 9.6 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.3493, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -1.202, 95% CI 2-sided [-3.729 to 1.324]
Statistical Analysis 2: Comparison: 3.2 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.0162, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -3.136, 95% CI 2-sided [-5.685 to -0.586]

2. Primary Outcome: Obsessive and Compulsive Behaviors
Description: Change in obsessive and compulsive behaviors as measured by the Children's Yale-Brown Obsessive-Compulsive Scale (CY-BOCS) Total Score versus placebo.
  Score range: 0-40; higher scores mean a worse outcome. Reduction in score indicates improvement.
Time Frame: baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Number analyzed (Participants) | 40 | 39 | 40
score on a scale | -2.968 [-4.667 to -1.268] | -3.123 [-4.843 to -1.403] | -2.360 [-4.046 to -0.674]
Statistical Analysis 1: Comparison: 9.6 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.6001, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -0.608, 95% CI 2-sided [-2.890 to 1.674]
Statistical Analysis 2: Comparison: 3.2 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.5143, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -0.764, 95% CI 2-sided [-3.068 to 1.541]

3. Secondary Outcome: Anxiety
Description: Change in participant anxiety as measured by the PWS Anxiety and Distress Questionnaire (PADQ) Total Score versus placebo.
  Score range: 0-56; higher scores mean a worse outcome. Reduction in score indicates improvement.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Number analyzed (Participants) | 40 | 39 | 40
score on a scale | -4.306 [-6.797 to -1.815] | -8.301 [-10.790 to -5.811] | -4.489 [-6.942 to -2.037]
Statistical Analysis 1: Comparison: 9.6 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.9144, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = 0.183, 95% CI 2-sided [-3.175 to 3.541]
Statistical Analysis 2: Comparison: 3.2 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.0266, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -3.812, 95% CI 2-sided [-7.177 to -0.446]

4. Secondary Outcome: Global Impression
Description: Clinical Global Impression of Change (CGI-C) score versus placebo. Score range: 1-7; higher scores mean a worse outcome. Reduction in score indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Number analyzed (Participants) | 40 | 39 | 40
score on a scale | 3.582 [3.250 to 3.913] | 3.395 [3.057 to 3.733] | 3.893 [3.562 to 4.225]
Statistical Analysis 1: Comparison: 9.6 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.1598, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -0.312, 95% CI 2-sided [-0.748 to 0.125]
Statistical Analysis 2: Comparison: 3.2 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.0266, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -0.498, 95% CI 2-sided [-0.937 to -0.059]

5. Secondary Outcome: Hyperphagia Behavior (Subset)
Description: Change in hyperphagia as measured by the change in specified subsets of HQ-CT questions versus placebo.
  Score range: 0-24; higher scores mean a worse outcome. Reduction in score indicates improvement.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
Number analyzed (Participants) | 40 | 39 | 40
score on a scale | -3.295 [-4.667 to -1.922] | -4.621 [-6.010 to -3.233] | -2.209 [-3.577 to -0.841]
Statistical Analysis 1: Comparison: 9.6 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.2479, Mixed Models Analysis — 0.05 threshold for statistical significance; Mean Difference (Net) = -1.085, 95% CI 2-sided [-2.932 to 0.761]
Statistical Analysis 2: Comparison: 3.2 mg of LV-101 vs Placebo; Test type: Superiority; p = 0.0114, Mixed Models Analysis — 0.05 for statistical significance; Mean Difference (Net) = -2.412, 95% CI 2-sided [-4.276 to -0.548]

ADVERSE EVENTS:
Time Frame: 8-week placebo-controlled period
Groups:
- 9.6 mg of LV-101: 9.6 mg of LV-101 during the 8-week placebo controlled period
  9.6 mg intranasal carbetocin: three times per day with meals
- 3.2 mg of LV-101: 3.2 mg of LV-101 during the 8-weeks placebo-controlled period
  3.2 mg intranasal carbetocin: three times per day with meals
- Placebo: Matched intranasal placebo during 8-week placebo-controlled period
  placebo: three times per day with meals
Arm/Group | 9.6 mg of LV-101 | 3.2 mg of LV-101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 20/44 | 19/43 | 10/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9.6 mg of LV-101 (N=44) | 3.2 mg of LV-101 (N=43) | Placebo (N=43)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (General disorders) | 2 (2) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 7 (8) | 3 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (2) | 1 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Flushing (Vascular disorders) | 9 (10) | 6 (6) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic began affecting this study in early March 2020 by substantially impacting the ability to safely enroll clinical study subjects, by requiring remote visits and monitoring, and by dramatically changing daily routines and social environments in this sensitive PWS population. Levo held new screening and enrollment in March 2020, and subsequently closed screening and enrollment in May 2020, resulting in the enrollment of 130 subjects instead of the 175 subjects planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study is a multi-center study. Sponsor retains first publication rights for a period of time after conclusion of study. Study has not yet completed.

DOCUMENTS (2):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03649477/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03649477/SAP_001.pdf